CLINICAL TRIAL: NCT01450748
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of Alginos Oral Suspension (Sodium Alginate 50 mg/ml) for the Treatment of Patients With Laryngopharyngeal Reflux (LPR)
Brief Title: Efficacy and Safety of Alginos Oral Suspension to Treat Laryngopharyngeal Reflux
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTYALG1101; NTUH-IRB-201106058MA (Other: TTY)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Laryngopharyngeal Reflux
Keywords: sodium alginate; laryngopharyngeal reflux; combined impedance-pH monitoring
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — Alginates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium alginate (Experimental): oral suspension, 50 mg/ml
  Interventions: Drug: Sodium alginate
- Placebo (Placebo Comparator): oral suspension without active ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium alginate — oral suspension, 50 mg/ml, 20 ml three times daily, 8 weeks
  Other Names: Alginos
  Arms: Sodium alginate
Drug: Placebo — matching placebo oral suspension, 50 mg/ml, 20 ml three times daily, 8 weeks
  Arms: Placebo

SUMMARY:
Laryngopharyngeal reflux (LPR), the backflow of gastric acid into the larynx and hypopharynx, is a contributing factor to hoarseness, throat clearing, throat pain, and globus sensation. The therapeutic effect of proton pump inhibitors (PPIs) is controversial because a high placebo effect can be observed. Sodium Alginate is an effective medication indicated for symptomatic treatment of gastroesophageal reflux. This randomized, double-blind, placebo-controlled study aims to evaluate the efficacy and safety profile of sodium alginates oral suspension (50 mg/ml) 20 ml 3 times daily for the treatment of with LPR patients in Taiwan. Efficacy assessments include mean reduction in the total reflux symptom index (RSI) score after 4 and 8 weeks treatment, mean reduction in the total reflux finding score (RFS) after 4 and 8 weeks treatment, mean changes in the total numbers of reflux episodes as measured by 24-hour ambulatory combined impedance-pH monitoring after 1 day and 8 weeks treatment. Safety assessments include incidence of adverse events. The study hypothesis is sodium alginate is superior over placebo in relieving LPR symptoms.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled trial aims to evaluate the efficacy and safety profiles of sodium alginate oral suspension (50mg/ml) 20ml 3 times daily for the treatment of patients with laryngopharyngeal reflux (LPR) in Taiwan. Patients will be enrolled into study if they are at the age of 12 to 75 years old, have at least one symptom consistent with LPR and lasting for more than 4 weeks before study, with a total reflux symptom index (RSI)>10, with a total reflux finding score (RFS)>5, and have signed the informed consent form. Patients will be excluded if they are diagnosed as erosive gastroesophageal reflux disease (GERD)as evidenced by upper GI endoscopy, viral or bacterial laryngitis, or occupational exposures causing laryngitis, laryngeal or hypopharyngeal cancer, esophageal or gastric cancer, with history of neck radiation therapy, with history of esophageal or gastric surgery, with active pulmonary infection (pneumonia, tuberculosis) as evidenced by chest X-ray, with endotracheal tube intubation within 2 months before entering study, or taking any alginate preparations within 2 days; H2-blocker, prokinetic agent or antacid within 7 days; or proton pump inhibitors (PPIs) within 14 days before screening. The primary efficacy endpoint is mean reduction in the total RSI from baseline to Week 8. The secondary efficacy endpoints are mean reduction in the total RSI from baseline to Day 2 and Week 4; mean reduction in the RFS from baseline to Week 4 and Week 8; mean change in the individual component of RSI from baseline to Day 2 , Week 4 and Week 8; mean change in the individual component of RFS from baseline to Week 4 and Week 8; and mean change in the total numbers of reflux episodes as measured by 24-hr ambulatory combined impedance-pH monitoring from baseline to day 2 and week 8. The safety endpoint is incidence of adverse events. The study hypothesis is that sodium alginate is superior over placebo in treating patients with LPR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of 12-75 years old (inclusive)
* Patients with at least one symptom consistent with LPR, including hoarseness, throat clearing, throat pain, globus sensation in the throat, or chronic cough ≧ 4 weeks before entering study
* Patients with a total reflux symptom index (RSI) >10 (based on a self-administered 9-item questionnaire of voice/throat complaints)
* Patients with a total reflux finding score (RFS) >5 (based on a laryngoscopic examination by investigators)
* Patients or their legal representatives have signed the informed consent form

Exclusion Criteria:

* Patients with viral or bacterial laryngitis, or occupational exposures causing laryngitis
* Patients with erosive GERD as evidenced by upper GI endoscopy
* Patients with laryngeal or hypopharyngeal cancer, esophageal or gastric cancer, , or with history of neck radiation therapy
* Patients with history of uncontrolled hypertension or moderate to severe renal impairment
* Patients with history of esophageal or gastric surgery
* Patients with active pulmonary infection (pneumonia, tuberculosis) as evidenced by chest X-ray
* Patients with endotracheal tube intubation within 2 months before entering study
* Patients had taken any alginate preparations within 2 days; H2-blocker, prokinetic agent or antacid within 7 days; or proton pump inhibitors (PPIs) within 14 days before screening
* Patients with a history of allergy to the study drugs or their related compounds
* Patients with a history of alcohol or drug abuse, or with any psychiatric disease
* Patients participated any investigational drug trial within 4 weeks before entering the study
* Patients with any other conditions or diseases that investigator considers it is not appropriate to enter the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean reduction in the total reflux symptom index (RSI) score from baseline to Week 8 | before and after 8 weeks treatment
  RSI is a self-administered 9-item questionnaire. RSI can be completed in less than 1 minute. The scale for each individual item ranges from 0 (no problem) to 5 (severe problem), with a maximum total score of 45. A total RSI score of >10 is suggestive of laryngopharyngeal reflux

SECONDARY OUTCOMES:
Mean reduction in the total reflux symptom index (RSI) score from baseline to Day 2 and Week 4 | before and after 1 day and 4 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yu Hsiao, Ph.D., Principal Investigator — Department of Ear, Nose and Throat, National Taiwan University Hospital
Locations (1):
- TTY Biopharm Company Limited Taipei Branch, Taipei, Taiwan